CLINICAL TRIAL: NCT01950845
Title: Per Operative Fluid Optimisation Comparison of an Automated Closed-Loop System Versus Current Practice in High Risk Abdominal Surgical Patient. A Prospective, Randomized Clinical Trial.
Brief Title: Automated Versus Manual Fluid Management for High Risk Abdominal Surgical Patient. A Prospective, Randomized Trial
Acronym: CL vs CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2012.770
Record Dates: First submitted 2013-09-17; First posted 2013-09-26 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Major Abdominal Surgery; Colorectal Surgery; Hepatectomy; Pancreatectomy; Pancreaticoduodenectomy
Keywords: anesthesiology, Closed-Loop system, automated fluid management, cardiac output optimization, high risk surgical patient, major abdominal surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Automated fluid management system (Closed-loop system) (Experimental): cardiac output Vigileo® (Edwards Lifesciences) monitoring is connected to the closed loop system that will automatically provide per operative fluid bolus to optimize cardiac output by automated detection of fluid responsiveness state.
  Interventions: Device: Closed loop automated System (LIR®: learning intravenous resuscitator)
- Current practice manual fluid management (Sham Comparator): cardiac output Vigileo® (Edwards Lifesciences) monitoring will be used to help the anesthesiologist team to detect fluid responsiveness state for the manual fluid management optimization
  Interventions: Device: manual current practice by anesthesiologist team

INTERVENTIONS:
Device: Closed loop automated System (LIR®: learning intravenous resuscitator) — Connection of the system to the patient under supervision of the anesthesiologist team during all the anesthesia procedure, respective of the applicability criteria for the fluid responsiveness detection.
  Arms: Automated fluid management system (Closed-loop system)
Device: manual current practice by anesthesiologist team — The anesthesiologist team will manage the fluid administration during all the anesthesia procedure.
  Arms: Current practice manual fluid management

SUMMARY:
Dynamic parameters like pulse pressure variation have been shown to be accurate predictors of fluid responsiveness. Hemodynamic optimization based on fluid management and stroke volume optimization have been shown to improve patient outcomes, especially for moderate and high risk abdominal surgical patients. A novel closed-loop fluid administration system based on multi-parameter hemodynamic monitoring have been described recently. This prospective, randomized, surgeon and patient blinded study aims at comparing the cardiac output provided by either this closed-loop system or the anesthesiologist team in high-rish surgical patient elected for abdominal surgery at Pierre Bénite University Hospital, Hospices Civils of Lyon, France. Primary endpoint is the mean indexed cardiac output during surgery per group. We will also compare hemodynamic parameter (cardiac output, stroke volume, blood pressure heart rate…) and patient's outcomes (morbidity, mortality, transfusion rate, hospital length of stay) between groups

ELIGIBILITY:
Inclusion Criteria:

* Elective major abdominal surgery
* Patient physical status ASA 2-4
* General anesthesia with positive pressure ventilation
* High risk surgical patient with a per operative Vigileo® cardiac output monitoring decided a priori.

Exclusion Criteria:

* Pregnant female
* Intraoperative hyperthermic chemotherapy procedure
* Patient physical status ASA more than 4
* Patient with allergy to hydroxyethyl starch
* Cardiac arrhythmia
* ventilation with tidal volume inferior 7mL/Kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Mean indexed cardiac output | J1 to J12 (Within the surgical hospital length of stay)

SECONDARY OUTCOMES:
per operative hemodynamic parameter | J1 (per operative time)
Per operative fluid administration | J1 (per operative)
Hospital length of stay | J1 to J12
  Within the surgical hospital length of stay
Occurrence of a adverse event after surgery | an expected average of 12 days
  Within the surgical hospital length of stay
Occurrence of a death whatever the cause | an expected average of 12 days
  Within the surgical hospital length of stay

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Lyon Sud, Hospices Civils de Lyon, Pierre-Bénite, France

REFERENCES:
- [Background] Lilot M, Bellon A, Gueugnon M, Laplace MC, Baffeleuf B, Hacquard P, Barthomeuf F, Parent C, Tran T, Soubirou JL, Robinson P, Bouvet L, Vassal O, Lehot JJ, Piriou V. Comparison of cardiac output optimization with an automated closed-loop goal-directed fluid therapy versus non standardized manual fluid administration during elective abdominal surgery: first prospective randomized controlled trial. J Clin Monit Comput. 2018 Dec;32(6):993-1003. doi: 10.1007/s10877-018-0106-7. Epub 2018 Jan 27. PMID 29380190